CLINICAL TRIAL: NCT05397509
Title: Effect of the Olive Leaf Tea Ingestion in Post-prandial Glycemic Response (OLIFTEA)
Acronym: OLIFTEA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Politécnico de Bragança (Other)
Responsible Party: Principal Investigator, Manuela Meireles, Researcher, Instituto Politécnico de Bragança
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 361221
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-04

CONDITIONS: Blood Glucose

STUDY DESIGN:
Intervention Model Description: Each participant will test one beverage on the first visit and the other one on the second visit. A wash-out period of two weeks will be done.
  Allocation of the first beverage to each participant is made by randomization.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: olive leaf tea and placebo tea were offered in a opaque mug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olive Leaf Tea (Experimental): Olive Leaf Tea
  Interventions: Other: Olive leaf tea
- Placebo tea (Placebo Comparator): Placebo tea
  Interventions: Other: Placebo tea

INTERVENTIONS:
Other: Olive leaf tea — 250 mL of Olive leaf tea and a high-glycemic breakfast
  Arms: Olive Leaf Tea
Other: Placebo tea — 250 mL of placebo tea and a high-glycemic breakfast
  Arms: Placebo tea

SUMMARY:
This study tests the effect of Olive Tea Ingestion in ameliorating glycemic response after a high-glycemic meal

DETAILED DESCRIPTION:
This study is a double-blinded, randomized, placebo-controlled clinical trial with cross-over design.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* currently taking drugs interfering with glucose regulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 50 female- 50 male
Enrollment: 20 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | 120 minutes
  Area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Meireles, PhD, Principal Investigator — Instituto Politécnico de Bragança
Locations (1):
- escola Superior de Saúde, Bragança, Portugal